CLINICAL TRIAL: NCT06995911
Title: A Randomized Controlled Clinical Trial on the Efficacy and Safety of the Virtual Far-sight Reading Device for Myopia Intervention in Pre-myopic Children
Brief Title: Virtual Far-sight Reading Device for Myopia Intervention Among Pre-myopic Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: YMZSSJLY202501
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Myopia; Pre-myopia
Keywords: Myopia; Pre-myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: This randomized controlled crossover trial was conducted in two sequential phases:
  Phase I (Day 0-90):
  Group A: Performed daily near-work activities (e.g., reading/writing) using the Virtual Far-sight Reading Device with cumulative daily use ≥60 minutes.
  Group B: Engaged in routine near-work activities without intervention.
  Phase II (Day 90-180):
  Group A: Switched to standard near-work practice without device use.
  Group B: Initiated Virtual Far-sight Reading Device intervention under identical protocol (≥60 min/day cumulative use).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nearwork with the Virtual Far-sight Reading Device (Experimental)
  Interventions: Device: Virtual Far-sight Reading Device
- Nearwork without the Virtual Far-sight Reading Device (No Intervention)

INTERVENTIONS:
Device: Virtual Far-sight Reading Device — The Virtual Far-sight Reading Device utilizes a birdbath optical configuration and freeform surface technology to extend the working distance from 30 cm to over 6 meters, thereby simulating distance viewing conditions and maintaining ciliary muscle relaxation. Study participants were required to engage in reading and writing tasks using the device for a cumulative daily duration of at least 1 hour.
  Arms: Nearwork with the Virtual Far-sight Reading Device

SUMMARY:
This clinical trial wants to find out if the Virtual Far-sight Reading Device can help prevent or slow down myopia progression in children and teenagers with pre-myopia. We also want to know what makes this treatment work better for some participants and check for any eye or body-related side effects over time.

Main questions:

Can using the Virtual Far-sight Reading Device reduce the risk of myopia? Is the device safe to use every day for up to 6 months?

What we'll do:

Researchers will compare two groups of children:

Group A: Uses the device for reading/writing (at least 1 hour daily) Group B: Does regular reading/writing without the device After 90 days, the groups will switch to see if the results stay the same.

Participants will:

* Have free eye checkups 3 times over 6 months
* Use the device during homework time (if in the desk group)
* Report any eye discomfort or problems

DETAILED DESCRIPTION:
The Virtual Far-sight Reading Device is an innovative ocular protection device integrating advanced far-image optical technology, designed to alleviate asthenopia and prevent myopia progression by simulating a long-distance visual environment. Utilizing a birdbath optical configuration and freeform surface technology, it extends the working distance from 30 cm to over 6 meters, mimicking natural distance viewing to induce ciliary muscle relaxation. The device incorporates a cinematic-grade 2K true-color retinal display combined with a peripheral defocus optical design to generate hyperopic retinal shifts, thereby suppressing myopia development. Additional features include an embedded high-resolution AI camera, full-spectrum LED auxiliary lighting (CCT 5000K, CRI >90), and compatibility with extensive e-learning resources, making it suitable for diverse scenarios such as online classes, reading, and writing tasks.

This study employs a randomized controlled crossover trial to evaluate the efficacy and safety of the device in pre-myopic children and adolescents. Participants are divided into Groups A and B, with Phase I (Days 0-90) requiring Group A to perform daily near-work activities using the device for ≥60 minutes of cumulative daily use, while Group B follows conventional near-work practices without intervention. During Phase II (Days 91-180), the interventions are reversed between groups. Comprehensive ophthalmic evaluations are conducted at baseline, Day 90, and Day 180 to assess changes in spherical equivalent refraction (SER), axial length (AL), myopia incidence rate, binocular visual function parameters, and ocular morphological metrics, ensuring rigorous analysis of both therapeutic outcomes and safety profiles.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6-12 years (inclusive), gender unrestricted.

  * Worse eye cycloplegic spherical equivalent refraction (SER): -0.5 D < SER ≤ +0.75 D; Cylinder ≤ -1.5 D in both eyes; Interocular anisometropia ≤ 1.5 D ③ Visual acuity: Best-corrected visual acuity (BCVA) ≤ 0.1 logMAR in both eyes. ④ Family history: At least one parent with myopia.

    * Intraocular pressure (IOP): 10-21 mmHg in both eyes; Interocular IOP difference ≤ 5 mmHg

      ⑥ Compliance: Commitment to daily home use of the Far-Image Light Field Desk per protocol, immediate notification to investigators if unable to comply, and completion of scheduled follow-ups.

      ⑦ Informed consent: Signed assent form (minor) and written informed consent from legal guardian.

Exclusion Criteria:

* Ocular comorbidities affecting vision/refractive development: Marfan syndrome; Lens pathologies (e.g., cataracts); Glaucoma; retinal detachment; retinopathy of prematurity

  * Systemic diseases: Immune/CNS disorders; Down syndrome; Severe cardiopulmonary/hepatic/renal dysfunction; Uncontrolled asthma

    * Ocular abnormalities: Manifest strabismus; Binocular vision dysfunction; Pathological ocular changes or active ocular inflammation ④ Recent myopia interventions (within 3 months prior to screening): Orthokeratology; multifocal contact lenses; Functional spectacles, red-light therapy

      ⑤ Medications affecting efficacy evaluation (within 3 months): Anticholinergics (e.g., atropine, pirenzepine); Cholinergics (e.g., pilocarpine)

      ⑥ Participation in other clinical trials within 3 months.

      ⑦ Contraindications/allergies to cycloplegics or study-related medications.

      ⑧ Chronic psychiatric disorders or cognitive impairment.

      ⑨ Other conditions deemed unsuitable by investigators.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Spherical Equivalent Refraction | 90 and 180 days from baseline

SECONDARY OUTCOMES:
Changes in Axial Length | 90 and 180 days from baseline
Cumulative Incidence of Myopia | 90 and 180 days from baseline

OTHER OUTCOMES:
Changes in Accommodative Response | 90 and 180 days from baseline
Changes in Facility of Accommodation | 90 and 180 days from baseline
Changes in Positive/Negative Relative Accommodation | 90 and 180 days from baseline
Changes in Amplitude of Accommodation | 90 and 180 days from baseline
Changes in Lens Thickness | 90 and 180 days from baseline
Changes in Choroidal Thickness | 90 and 180 days from baseline
Changes in Best Corrected Visual Acuity | 90 and 180 days from baseline
Changes in Strabismus | 90 and 180 days from baseline
Changes in Asthenopia Score | 90 and 180 days from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Eye Disease Prevention and Treatment Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided